CLINICAL TRIAL: NCT01878487
Title: INtra-Vascular Ultrasound Study of Export Thrombectomy in ST Elevation Myocardial Infarction Myocardial Infarction
Brief Title: Assessment of Lumen Expansion After Thrombus Extraction in Primary Percutaneous Coronary Intervention
Acronym: INVEST-MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0906/85
Record Dates: First submitted 2013-05-01; First posted 2013-06-17 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Acute ST Elevation Myocardial Infarction
Keywords: Acute MI; Primary percutaneous coronary intervention; thrombus aspiration, IVUS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Only one arm (Other): All patients will receive the same treatment, i.e. there is no randomization. There is therefore only one arm, all patients will by treated as per standard practice with thrombus aspiration and stenting as required, the lumen size of the vessel will be assessed with intravascular ultrasound at baseline, after thrombus aspiration and after stenting.
  Interventions: Device: Thrombus aspiration (Intravascular Ultrasound catheter (Boston))

INTERVENTIONS:
Device: Thrombus aspiration (Intravascular Ultrasound catheter (Boston)) — There is a single arm in the study where all patients are undergoing primary percutaneous coronary intervention for an acute myocardial infarction.
  All patients will have an Intravascular Ultrasound three times:
  1. At baseline
  2. After thrombus aspiration with a thrombus extraction catheter
  3. After stent deployment
  We are however assessing the physiological response of patients having an acute myocardial infarction and this is not a test of the devices as such.
  Other Names: Export thrombus aspiration cathether; Intravascular Ultrasound catheter (Boston)

SUMMARY:
To use IVUS to assess (1) culprit plaque morphology and thrombus burden in patients with ST-elevation myocardial infarction; (2) the efficacy of thrombus removal with an aspiration catheter in 40 patients during primary PCI.

DETAILED DESCRIPTION:
Primary PCI has become the preferred therapy for ST-elevation acute myocardial infarction. The TAPAS trial data suggests that widespread adoption of manual thrombus aspiration may improve clinical outcomes for patients undergoing primary PCI.

Little data exists on the degree to which thrombus is removed during thrombectomy and how much thrombus remains with the potential for distal embolisation during stent deployment. The mechanism of lumen enlargement after thrombus aspiration is also unknown. Since angiography only provides an outline image of the vascular lumen, such questions cannot be adequately addressed by this modality alone.

The aim of this study is to use IVUS to assess (1) culprit plaque morphology and thrombus burden in patients with ST-elevation myocardial infarction; (2) the efficacy of thrombus removal with an aspiration catheter during primary PCI.

Hypotheses In this study we will assess 40 patients with STEMI. Primary PCI will be performed according to our hospital standard working protocol with thrombus aspiration and balloon dilatation of the culprit lesion if necessary prior to stent deployment. IVUS imaging will be undertaken prior to, and following, passage of the aspirations catheter to assess (1) initial and (2) residual thrombus volume. A third and final IVUS imaging run will be performed after stenting of the culprit lesion. IVUS analysis will be performed off-line to assess the lumen enlargement and volume of residual thrombus at each stage. All studies will be undertaken with the approval of the local Clinical Research Ethics.

Aspirated material will be collected and analyzed. Clinical markers such as Troponin release and left ventricular function will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. patients 18-75 years old with myocardial infarction with ST-segment elevation
2. symptoms of myocardial ischemia lasting more than 30 minutes
3. onset of symptoms within 12 hours of hospital presentation
4. ST-segment elevation of more than 0.1 mV in two or more leads on the ECG

Exclusion Criteria:

1. inability to obtain informed consent
2. use of fibrinolytic drug within 12 hours of presentation
3. comorbidity with anticipated life expectancy of < 6 months
4. cardiogenic shock on presentation
5. major bleeding diathesis
6. history of aspirin and clopidogrel intolerance
7. critical left main stem lesions
8. severe calcfic disease precluding safe passage of the imaging catheter
9. culprit lesion within saphenous vein grafts

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Coronary artery lumen expansion after thrombus aspiration in primary percutaneous intervention. | Day 1
  Degree of thrombus extraction can be visualised immediately by intravascular ultrasound (IVUS) but detailed analysis will be carried out off-line and by histopathology of aspirated material within 4 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Freeman Hospital, Newcastle, United Kingdom